CLINICAL TRIAL: NCT05415826
Title: Slow-Release Dexamethasone in Reducing Proliferative Vitreoretinopathy After Vitreotomy in Proliferative Diabetic Retinopathy
Brief Title: Ozurdex in Reducing PVR After Vitreotomy in PDR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PKUPHoph
Record Dates: First submitted 2022-06-08; First posted 2022-06-13 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Diabetic Retinopathy
Keywords: PDR; PVR; Ozurdex
MeSH Terms: conditions — Diabetic Retinopathy; Vitreoretinopathy, Proliferative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PPV group (Active Comparator): Eyes with proliferative diabetic retinopathy underwent PPV surgery with silicone oil filling.
  Interventions: Procedure: slow-release dexamethasone implant
- PPV+implant group (Experimental): Eyes with proliferative diabetic retinopathy underwent PPV surgery with silicone oil filling and slow-release dexamethasone implant.
  Interventions: Procedure: slow-release dexamethasone implant

INTERVENTIONS:
Procedure: slow-release dexamethasone implant — The eyes with proliferative diabetic retinopathy underwent PPV with silicone oil filling with or without slow-release dexamethasone implant at the end of surgery.

SUMMARY:
Diabetic retinopathy is a significant source of visual morbidity in the adult population. Complications of diabetic retinopathy include ischemic maculopathy, macular edema, and sequelae of fibrovascular proliferation, such as vitreous hemorrhage (VH), tractional retinal detachment (TRD), and neovascular glaucoma.Pars plana vitrectomy (PPV) is traditionally performed for nonclearing VH, significant fibrovascular proliferation, refractive macular edema, and/or TRD, particularly if macula-involving. However, the pathogenesis is complex and multifactorial: Pro-infammatory cytokines and chemokines signifcantly contribute to the disease development and promote ischemic changes in the retina. Therefore, there is a potential role for intravitreal steroids in disease modifcation.

DETAILED DESCRIPTION:
Diabetic retinopathy is a significant source of visual morbidity in the adult population. Complications of diabetic retinopathy include ischemic maculopathy, macular edema, and sequelae of fibrovascular proliferation, such as vitreous hemorrhage (VH), tractional retinal detachment (TRD), and neovascular glaucoma.Pars plana vitrectomy (PPV) is traditionally performed for nonclearing VH, significant fibrovascular proliferation, refractive macular edema, and/or TRD, particularly if macula-involving. However, the pathogenesis is complex and multifactorial: Pro-infammatory cytokines and chemokines signifcantly contribute to the disease development and promote ischemic changes in the retina. Therefore, there is a potential role for intravitreal steroids in disease modifcation. Corticosteroids reduce not only leukostasis and infammatory cytokine production, but also VEGF expression. Experimentally, corticosteroids potentially can influence both the inflammatory and the proliferative components of the PVR process via a variety of modes of administration without evidence of demonstrable retinal toxicity. So, this study is carried out for the purpose of investigating the efficacy of slow-release dexamethasone implant in proliferative vitreoretinopathy of postoperative proliferative diabetic retinopathy.

ELIGIBILITY:
Inclusion Criteria:

* macula off treatment naive TRD second to PDR causing visual loss;
* treated by standardize PPV, endolaser and silicone oil tamponade with or without DEX implant at the end of the surgery within 12 months from diagnosis of TRD;
* Hba1c is less than 10% with type 1 or 2 diabetes mellitus

Exclusion Criteria:

* other concomitant ocular diseases that cause RD ( for example rhegmatogenous retinal detachment, exudative retinal detachment, other causes for TRD);
* any previous injection of DEX implant;
* abnormalities of the vitreoretinal interface, such as epiretinal membrane, vitreomacular traction without RD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-15 (Estimated); Primary Completion 2022-09-15 (Estimated); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
PVR | during 3 months after surgery
  proliferative vitreoretinopathy after sugery
CRT | from preoperation to 3 months follow-up
  central retina thickness

SECONDARY OUTCOMES:
BCVA | from preoperation to 3 months follow-up
  best corrected visual acuity
Intraretinal hemorrhage | during 3 months after surgery
  Intraretinal hemorrhage

CONTACTS AND LOCATIONS:
Overall Officials: Jinfeng Qu, MD, Study Chair — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moss SE, Klein R, Klein BE. The 14-year incidence of visual loss in a diabetic population. Ophthalmology. 1998 Jun;105(6):998-1003. doi: 10.1016/S0161-6420(98)96025-0. PMID 9627648
- [Background] Fong DS, Ferris FL 3rd, Davis MD, Chew EY. Causes of severe visual loss in the early treatment diabetic retinopathy study: ETDRS report no. 24. Early Treatment Diabetic Retinopathy Study Research Group. Am J Ophthalmol. 1999 Feb;127(2):137-41. doi: 10.1016/s0002-9394(98)00309-2. PMID 10030553
- [Background] Early vitrectomy for severe vitreous hemorrhage in diabetic retinopathy. Four-year results of a randomized trial: Diabetic Retinopathy Vitrectomy Study Report 5. Arch Ophthalmol. 1990 Jul;108(7):958-64. doi: 10.1001/archopht.1990.01070090060040. PMID 2196036
- [Background] Vujosevic S, Simo R. Local and Systemic Inflammatory Biomarkers of Diabetic Retinopathy: An Integrative Approach. Invest Ophthalmol Vis Sci. 2017 May 1;58(6):BIO68-BIO75. doi: 10.1167/iovs.17-21769. PMID 28510630
- [Background] Funatsu H, Yamashita H, Noma H, Mimura T, Nakamura S, Sakata K, Hori S. Aqueous humor levels of cytokines are related to vitreous levels and progression of diabetic retinopathy in diabetic patients. Graefes Arch Clin Exp Ophthalmol. 2005 Jan;243(1):3-8. doi: 10.1007/s00417-004-0950-7. Epub 2004 Jul 17. PMID 15258777
- [Background] Schwartzman ML, Iserovich P, Gotlinger K, Bellner L, Dunn MW, Sartore M, Grazia Pertile M, Leonardi A, Sathe S, Beaton A, Trieu L, Sack R. Profile of lipid and protein autacoids in diabetic vitreous correlates with the progression of diabetic retinopathy. Diabetes. 2010 Jul;59(7):1780-8. doi: 10.2337/db10-0110. Epub 2010 Apr 27. PMID 20424229
- [Background] Goldberg RB. Cytokine and cytokine-like inflammation markers, endothelial dysfunction, and imbalanced coagulation in development of diabetes and its complications. J Clin Endocrinol Metab. 2009 Sep;94(9):3171-82. doi: 10.1210/jc.2008-2534. Epub 2009 Jun 9. PMID 19509100
- [Background] dell'Omo R, Semeraro F, Bamonte G, Cifariello F, Romano MR, Costagliola C. Vitreous mediators in retinal hypoxic diseases. Mediators Inflamm. 2013;2013:935301. doi: 10.1155/2013/935301. Epub 2013 Jan 10. PMID 23365490
- [Background] Albini TA, Abd-El-Barr MM, Carvounis PE, Iyer MN, Lakhanpal RR, Pennesi ME, Chevez-Barrios P, Wu SM, Holz ER. Long-term retinal toxicity of intravitreal commercially available preserved triamcinolone acetonide (Kenalog) in rabbit eyes. Invest Ophthalmol Vis Sci. 2007 Jan;48(1):390-5. doi: 10.1167/iovs.06-0145. PMID 17197559